CLINICAL TRIAL: NCT00760994
Title: Reducing Alcohol Use & PTSD w/ Cognitive Restructuring & Experiential Acceptance
Brief Title: Reducing Alcohol Use & Post-traumatic Stress Disorder (PTSD) With Cognitive Restructuring & Experiential Acceptance
Acronym: COPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); VA Puget Sound Health Care System (U.S. Federal Agency); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21AA017130-01 (NIH); R21AA017130 (NIH)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Alcoholism; Stress Disorders, Post-Traumatic
Keywords: Alcohol; Alcoholic; Alcoholism; Post-traumatic stress disorder; PTSD; Experiential acceptance; Mindfulness; Meditation; Meditate; Cognitive restructuring; Cognitive; Behavioral; Therapy; Treatment; Study; Intervention
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic; Behavior | interventions — Mindfulness; Cognitive Restructuring; Cognitive Behavioral Therapy; Food; Nutrition Policy; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 - Experiential Accepatance (Experimental): Experiential acceptance
  Interventions: Behavioral: Experiential acceptance
- 2 - Cognitive Restructuring (Active Comparator): Cognitive restructuring
  Interventions: Behavioral: Cognitive restructuring
- 3 - Control (Placebo Comparator): No-intervention control: Nutrition information
  Interventions: Other: No-intervention control: Nutrition information

INTERVENTIONS:
Behavioral: Experiential acceptance — The experiential acceptance coping condition will focus on changing one's relationship to one's internal events by learning to remain in contact with negative and positive thoughts and feelings and cravings as they are, without defense or judgment or attempting to cling to them (Eifert & Forsyth, 2005; Hayes, Strosahl, & Wilson, 1999; Kadden et al., 1992; Levitt, Brown, Orsillo, & Barlow, 2004).
  Other Names: Mindfulness meditation
  Arms: 1 - Experiential Accepatance
Behavioral: Cognitive restructuring — The cognitive restructuring coping condition will focus on how to change the content and frequency of internal events by changing one's thinking patterns (Kadden et al., 1992).
  Other Names: Cognitive-behavioral therapy
  Arms: 2 - Cognitive Restructuring
Other: No-intervention control: Nutrition information — The no-intervention condition will be taught the plate method, a nutritional servings guideline, which will have no content related to AUD or PTSD, in order to control for time and contact with a research assistant.
  Other Names: Plate method; Food; Nutrition guidelines; Diet
  Arms: 3 - Control

SUMMARY:
The purpose of this study is to determine whether an experiential acceptance therapy intervention is effective in the treatment of alcohol dependency and post-traumatic stress disorder (PTSD) symptoms in individuals who suffer from PTSD.

DETAILED DESCRIPTION:
Alcohol dependence (AD) afflicts nearly 14% of the population (Kessler et al., 1994; Kessler et al., 1997; Regier et al., 1990), and has a chronic and relapsing course (Brownell, Marlatt, Litchenstein, & Wilson, 1986). Negative emotional states have consistently been found to maintain alcohol use disorders (AUDs; Cooney, Litt, Morse, Bauer, & Gaupp, 1997; Litt, Cooney, Kadden, & Gaupp, 1990; Rubonis et al., 1994) and increase the risk of relapse following AUD treatment (Cooney et al., 1997). This relationship is particularly robust among individuals with co-morbid psychiatric disorders, such as posttraumatic stress disorder (PTSD; Coffey et al., 2002; Sharkansy, Brief, Peirce, Meehan, & Mannix, 1999; Tate, Brown, Unrod, & Ramo, 2004; Waldrop, Back, Verduin, & Brady, in press). Likewise, alcohol use may be maintained by a desire to facilitate or prolong positive emotional states (Cooper, Frone, Russell, & Mudar, 1992; Simpson, 2003).

Many psychological interventions for AUDs, most notably the majority of cognitive-behavioral treatment (CBT) packages, have thus focused on the development of coping skills to prevent relapse in response to such triggers, and have been demonstrated to be at least moderately effective in promoting abstinence (Miller & Wilbourne, 2002). However, attempts to specify the active ingredients of CBT for AD have been disappointing and most studies examining potential mechanisms of change have failed to find the expected relationships (Longabaugh et al., 2005; Morgenstern & Longabaugh, 2000). The lack of empirical evidence substantiating coping skills as a mechanism of change for CBT (Morgenstern & Longabaugh, 2000) may be due, in part, to the lack of specificity in coping skill interventions. Broadly speaking, two primary foci of coping skill interventions for AUD are 1) increasing cognitive techniques focused on challenging and changing thought patterns, or 2) increasing experiential acceptance by fostering an accepting stance towards internal states, such as through "urge surfing" (Kadden et al., 1992). These two coping skill approaches (cognitive restructuring and experiential acceptance) likely lead to reduced alcohol use through different pathways. Theoretically, experiential acceptance approaches suggest that the mechanism of change in decreasing alcohol use is increased willingness toward internal experience (e.g., emotions, thoughts, sensations), whereas cognitive restructuring approaches suggest that decreased alcohol use results from decreases in negative appraisals brought about by challenging and changing thought patterns. However, this has yet to be systematically evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years
* current DSM-IV diagnosis of alcohol dependence (AD) with some alcohol use in the last month
* current DSM-IV diagnosis of post-traumatic stress disorder (PTSD)
* capacity to provide informed consent
* English fluency
* no planned absences that they would be unable to complete 6 weeks of daily monitoring and study sessions
* access to a telephone
* desire to decrease or stop alcohol drinking behavior

Exclusion Criteria:

* a history of delirium tremens
* seizures, in order to ensure that participants will be medically safe to decrease alcohol use
* opiate abuse or dependence use or chronic treatment with any opioid- containing medications during the previous month
* currently taking or planning to start taking either antabuse or naltrexone (due to their pharmacological impact on alcohol cravings and use)
* exhibits signs or symptoms of alcohol withdrawal at the time of initial consent
* acutely suicidal with intent/plan or present an imminent danger to others
* a current psychotic disorder

For ethical reasons and because of the preliminary nature of this study, participants may be in ongoing substance abuse or mental health treatment (MH) or may initiate counseling or medications (other than those noted in exclusion criteria) during the course of the study. Mental health treatment involvement will be used as a covariate if it is related to study dependent variables.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy L Simpson, Ph.D., Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Background] Litt MD, Cooney NL, Kadden RM, Gaupp L. Reactivity to alcohol cues and induced moods in alcoholics. Addict Behav. 1990;15(2):137-46. doi: 10.1016/0306-4603(90)90017-r. PMID 2343787
- [Background] Brownell KD, Marlatt GA, Lichtenstein E, Wilson GT. Understanding and preventing relapse. Am Psychol. 1986 Jul;41(7):765-82. doi: 10.1037//0003-066x.41.7.765. No abstract available. PMID 3527003
- [Background] Cooney NL, Litt MD, Morse PA, Bauer LO, Gaupp L. Alcohol cue reactivity, negative-mood reactivity, and relapse in treated alcoholic men. J Abnorm Psychol. 1997 May;106(2):243-50. doi: 10.1037//0021-843x.106.2.243. PMID 9131844
- [Background] Coffey SF, Saladin ME, Drobes DJ, Brady KT, Dansky BS, Kilpatrick DG. Trauma and substance cue reactivity in individuals with comorbid posttraumatic stress disorder and cocaine or alcohol dependence. Drug Alcohol Depend. 2002 Jan 1;65(2):115-27. doi: 10.1016/s0376-8716(01)00157-0. PMID 11772473
- [Background] Cooper ML, Frone MR, Russell M, Mudar P. Drinking to regulate positive and negative emotions: a motivational model of alcohol use. J Pers Soc Psychol. 1995 Nov;69(5):990-1005. doi: 10.1037//0022-3514.69.5.990. PMID 7473043
- [Background] Kessler RC, McGonagle KA, Zhao S, Nelson CB, Hughes M, Eshleman S, Wittchen HU, Kendler KS. Lifetime and 12-month prevalence of DSM-III-R psychiatric disorders in the United States. Results from the National Comorbidity Survey. Arch Gen Psychiatry. 1994 Jan;51(1):8-19. doi: 10.1001/archpsyc.1994.03950010008002. PMID 8279933
- [Background] Kessler RC, Crum RM, Warner LA, Nelson CB, Schulenberg J, Anthony JC. Lifetime co-occurrence of DSM-III-R alcohol abuse and dependence with other psychiatric disorders in the National Comorbidity Survey. Arch Gen Psychiatry. 1997 Apr;54(4):313-21. doi: 10.1001/archpsyc.1997.01830160031005. PMID 9107147
- [Background] Longabaugh R, Donovan DM, Karno MP, McCrady BS, Morgenstern J, Tonigan JS. Active ingredients: how and why evidence-based alcohol behavioral treatment interventions work. Alcohol Clin Exp Res. 2005 Feb;29(2):235-47. doi: 10.1097/01.alc.0000153541.78005.1f. PMID 15714046
- [Background] Miller WR, Wilbourne PL. Mesa Grande: a methodological analysis of clinical trials of treatments for alcohol use disorders. Addiction. 2002 Mar;97(3):265-77. doi: 10.1046/j.1360-0443.2002.00019.x. PMID 11964100
- [Background] Morgenstern J, Longabaugh R. Cognitive-behavioral treatment for alcohol dependence: a review of evidence for its hypothesized mechanisms of action. Addiction. 2000 Oct;95(10):1475-90. doi: 10.1046/j.1360-0443.2000.951014753.x. PMID 11070524
- [Background] Regier DA, Farmer ME, Rae DS, Locke BZ, Keith SJ, Judd LL, Goodwin FK. Comorbidity of mental disorders with alcohol and other drug abuse. Results from the Epidemiologic Catchment Area (ECA) Study. JAMA. 1990 Nov 21;264(19):2511-8. PMID 2232018
- [Background] Rubonis AV, Colby SM, Monti PM, Rohsenow DJ, Gulliver SB, Sirota AD. Alcohol cue reactivity and mood induction in male and female alcoholics. J Stud Alcohol. 1994 Jul;55(4):487-94. doi: 10.15288/jsa.1994.55.487. PMID 7934057
- [Background] Simpson TL. Childhood sexual abuse, PTSD, and the functional roles of alcohol use among women drinkers. Subst Use Misuse. 2003 Jan;38(2):249-70. doi: 10.1081/ja-120017248. PMID 12625430
- [Background] Tate SR, Brown SA, Unrod M, Ramo DE. Context of relapse for substance-dependent adults with and without comorbid psychiatric disorders. Addict Behav. 2004 Dec;29(9):1707-24. doi: 10.1016/j.addbeh.2004.03.037. PMID 15530716
- [Background] Eifert, G.H., & Forsyth, J.P. (2005) Acceptance & commitment therapy for anxiety disorders: A practitioner's treatment guide to using mindfulness, acceptance, and values-based behavior change strategies. Oakland, CA: New Harbinger Publications.
- [Background] Hayes, S. C., Strosahl, K. D., & Wilson, K. G. (1999). Acceptance and commitment therapy: An experiential approach to behavior change. New York: Guilford Press.
- [Background] Kadden, R. M., Carroll, K., Donovan, D., Cooney, N. L., Monti, P., Abrams, D., et al. (1992). Cognitive-behavioral coping skills therapy manual: A clinical research guide for therapists treating individuals with alcohol abuse and dependence (Vol. 3; Project MATCH Monograph, DHHS Publication No 92-1895). Washington, DC: U. S. Government Printing Office.
- [Background] Levitt, J. T., Brown, T. A., Orsillo, S. M., & Barlow, D. H. (2004). The effects of acceptance versus suppression of emotion on subjective and psychophysiological response to carbon dioxide challenge in patients with panic disorder. Behavior Therapy, 35, 747-766.
- [Background] Sharkansky, E. J., Brief, D. P., Peirce, J. M., Meehan, J. C., & Mannix, L. M. (1999). Substance abuse patients with posttraumatic stress disorder (PTSD): Identifying specific triggers of substance use and their associations with PTSD symptoms. Psychology of Addictive Behaviors, 13, 89-97.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant who wanted to decrease their alcohol use were recruited through newspaper advertisements & flyers. One hundred thirty two individuals were consented, 92 out of the 132 consented individuals were eligible, and 80 were randomized. Seventy eight participants received an intervention.
Pre-assignment Details: Out of 132 individuals who provided written consent, 40 were ineligible:
  1. 10 individuals didn't use alcohol or have an alcohol diagnosis.
  2. 16 individuals didn't have PTSD.
  3. 4 individuals used an opiate or methamphetamine.
  4. 7 individuals had a bipolar disorder or psychotic.
  5. 3 individuals had reasons other than the ones above.
Groups:
- 1 - Experiential Accepatance (EA): Experiential acceptance
  Experiential acceptance: The experiential acceptance coping condition will focus on changing one's relationship to one's internal events by learning to remain in contact with negative and positive thoughts and feelings and cravings as they are, without defense or judgment or attempting to cling to them (Eifert & Forsyth, 2005; Hayes, Strosahl, & Wilson, 1999; Kadden et al., 1992; Levitt, Brown, Orsillo, & Barlow, 2004).
- 2 - Cognitive Restructuring (CR): Cognitive restructuring
  Cognitive restructuring: The cognitive restructuring coping condition will focus on how to change the content and frequency of internal events by changing one's thinking patterns (Kadden et al., 1992).
Period: Overall Study
Arm/Group | 1 - Experiential Accepatance (EA) | 2 - Cognitive Restructuring (CR) | 3 - Control
Started | 29 | 31 | 20
Completed | 25 | 27 | 17
Not Completed | 4 | 4 | 3
Not completed — Lost to Follow-up | 4 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Two of the 29 participants in the Experiential Acceptance group didn't receive the intervention, thus their data weren't included in the baseline and outcome analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Experiential Accepatance (EA) | 2 - Cognitive Restructuring (CR) | 3 - Control | Total
Number analyzed (Participants) | 27 | 31 | 20 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.93 (12.34) | 42.97 (12.44) | 46.95 (8.75) | 44.32 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 10 | 38
  Male | 15 | 15 | 10 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 11 | 11 | 12 | 34
  Asian | 0 | 1 | 0 | 1
  Hispanic | 2 | 1 | 0 | 3
  Native American | 1 | 0 | 1 | 2
  White (non Hispanic) | 10 | 16 | 7 | 33
  Multiple race | 1 | 1 | 0 | 2
  Other | 2 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 31 | 20 | 78
Average Drinks per Day Assessed Using Daily Interactive Voice Response (IVR) [Mean (Standard Deviation); unit: drinks per day] — One week prior to treatment, participants reported their alcohol use on the previous day using the IVR technology. Each participant's data were added and averaged to get the baseline average drinks per day of each treatment group (EA and CR) and control group. The higher the number, the more drinks were consumed per day. Possible minimum value: 0. Possible maximum value: unlimited.
  drinks per day | 5.2 (5.9) | 2.7 (3.5) | 4.6 (4.7) | 4.0 (4.8)
Average PTSD Scores per Day Assessed Using Daily Interactive Voice Response (IVR) [Mean (Standard Deviation); unit: units on a scale] — One week prior to treatment, participants completed an abbreviated version of PCL-C (PTSD Checklist-Civilian Version) daily via the IVR technology. Three re-experiencing symptoms, 2 avoidance symptoms, 3 emotional numbing symptoms, & 4 four hyperarousal symptoms were included. Participants rated each symptom from 0 (not at all) to 8 (all the time). The higher the score, the more intense their PTSD symptoms. The minimum & maximum possible scores were 0 & 96, respectively. Each participant's data were added and averaged to get the average baseline PTSD scores per day for each group.
  units on a scale | 3.2 (1.6) | 3.9 (1.6) | 4.0 (1.4) | 3.7 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Average Drinks Per Day Assessed Using Daily Interactive Voice Response (IVR)
Description: After the treatment had been started and for five weeks following the treatment, participants reported their alcohol use on the previous day using the IVR technology. Each participant's data were added and averaged to get the average drinks per day of each treatment group (EA and CR) and control group. The higher the number, the more drinks were consumed per day. Possible minimum value: 0. Possible maximum value: unlimited.
Time Frame: 5 weeks
Population: Data were analyzed using Generalized Estimating Equation (GEE) models.
Measure: Mean (Standard Deviation); unit: drinks per day
Arm/Group | 1 - Experiential Accepatance | 2 - Cognitive Restructuring | 3 - Control
Number analyzed (Participants) | 27 | 31 | 20
drinks per day | 3.6 (5) | 1.8 (2.5) | 3.1 (3.7)

2. Secondary Outcome: Average Post-Traumatic Stress Disorder (PTSD) Scores Per Day Assessed Using Daily Interactive Voice Response (IVR)
Description: PTSD scores were collected via the IVR technology after the treatment has been started and for the next five weeks. Participants completed an abbreviated version of PCL-C (PTSD Checklist-Civilian Version) daily. Three re-experiencing symptoms, 2 avoidance symptoms, 3 emotional numbing symptoms, & 4 four hyperarousal symptoms were included. Participants rated each symptom from 0 (not at all) to 8 (all the time). The higher the score, the more intense their PTSD symptoms. The minimum & maximum possible scores were 0 & 96, respectively. Each participant's data were added and averaged to get the average PTSD scores per day of each treatment group (EA and CR) and control group.
Time Frame: 5 weeks
Population: Data were analyzed using Generalized Estimating Equation (GEE) models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 - Experiential Accepatance (EA) | 2 - Cognitive Restructuring (CR) | 3 - Control
Number analyzed (Participants) | 27 | 31 | 20
units on a scale | 2.7 (1.4) | 3.1 (1.8) | 3.0 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected on the average of 44 days/participant, with a range of 42 to 71 days. Our first participant joined the study in May 2009 and the last participant completed the study in December 2010 (1 year and 7 months).
Description: We did not systematically collect adverse events, but participants had opportunities to report adverse events throughout follow-up calls and in-person visits.
Arm/Group | 1 - Experiential Accepatance (EA) | 2 - Cognitive Restructuring (CR) | 3 - Control
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/31 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/31 | 0/20
Other Adverse Events (participants affected / at risk) | 0/27 | 0/31 | 0/20

LIMITATIONS AND CAVEATS:
Limitations of the present study:

1. The study had a short follow-up assessment period (5 weeks) & did not assess all PTSD symptoms.

3. Asking participants to recall & report drinking on a daily basis may have enhanced the impacts of interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2010-12-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT00760994/ICF_000.pdf